CLINICAL TRIAL: NCT01319994
Title: Prevention of Metabolic Complications of Glucocorticoid Excess - a Randomised, Doubleblind,Placebo Controlled Study
Brief Title: Prevention of Metabolic Complications of Glucocorticoid Excess
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Barts and the London School of Medicine and Dentistry (Other)
Responsible Party: Principal Investigator, Marta Korbonits, Professor, Barts & The London NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09/H1102/82
Record Dates: First submitted 2011-02-21; First posted 2011-03-22 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-01

CONDITIONS: Iatrogenic Cushing Disease
Keywords: glucocorticoid
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): Metformin 850mg TDS (12 weeks)
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo 850mg TDS (12 weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin 850mg TDS (12 weeks)
  Other Names: metformin tablet containing 850mg metformin
  Arms: Metformin
Drug: Placebo — Placebo 850mg TDS (12 weeks)
  Other Names: Placebo tablet matching the active drug tablet
  Arms: Placebo

SUMMARY:
According to current estimates, nearly 1% of the general population is treated with long-term glucocorticoids. Chronic hypercortisolism leads to a phenotype that resembles the metabolic syndrome. The investigators have shown that inhibition of adenosine-monophosphate-activated protein kinase (AMPK) activity in adipose tissue plays a role in corticosteroid-mediated insulin resistance. Metformin, one of the mainstay therapies for type 2 diabetes, is a known activator of AMPK, which mediates its beneficial effects on glucose and lipid metabolism. The investigators have shown in an animal model that metformin - via altering AMPK activity - prevents the development of the metabolic complications of glucocorticoid excess, and the investigators wish to confirm this in a human study. The aim of this prospective, randomised, double-blind, placebo-controlled study is to investigate the effect of metformin treatment on metabolic parameters in patients on long-term high-dose glucocorticoids. The study is part of the investigators translational project and could rapidly lead to immediate patient benefit, improving quality of life and reducing health care costs for the NHS.

DETAILED DESCRIPTION:
2 Study Aims and Objectives To investigate the effect of metformin treatment on metabolic parameters in patients with long-term high dose GCs.

3 Study Design 3.1 General Design We will recruit patients (18-75y) requiring glucocorticoid treatment for various inflammatory conditions (e.g. rheumatoid arthritis, giant cell arteritis/polymyalgia rheumatic, asthma, sarcoidosis) into a pilot, randomised, double-blind, placebo-controlled trial. These patients will be treated with metformin to prevent or reverse their metabolic complications. Prevention algorithm: Patients who are about to start GC treatment predictably for ≥12w at a ≥10mg/d prednisolone (or equivalent) dose who consent to participate in this study will be randomly assigned to receive either placebo (20 patients/group, see power calculations) or metformin at the maximum tolerated dose with a minimum of 850 mg bd for 12w. Treatment algorithm: Consenting patients already on long-term GC treatment (≥4w, ≥20mg/d prednisolone or equivalent) who are expected to continue for at least 12w at ≥10mg/d prednisolone will be randomly assigned to receive either placebo or metformin for 12w. In both algorithms, metformin treatment will be started gradually (as standard practice) to avoid gastrointestinal side effects and the full dose will be reached by day 10. Patients will have a full clinical assessment before the start of the metformin treatment and at the end of the 12w treatment period. Anthropometric and biochemical parameters and questionnaires will be repeated at 4 and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with an inflammatory condition and not started yet on GC treatment or • patients with an inflammatory condition treated with GC >20mg/d of prednisolone (or its cumulative equivalent) for at least 4wks
* minimal duration of prospective therapy 12w
* dose of prednisolone ≥10mg/d (or equivalent GC)
* ambulatory patients
* patients >18 years old
* ability to understand verbal and written instructions and informed consent

Exclusion Criteria:

* prior therapy with metformin during the last 6 months
* known pre-existing diabetes
* pregnancy
* breastfeeding
* liver impairment: ALT and/or AST ≥2.5 x UNL
* renal impairment: serum creatinine levels ≥135.0 µmol/L in males and ≥110.0 µmol/L in females
* current malignancy
* patients unable to give written informed consent
* or patients not understanding English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-07; Primary Completion 2014-08 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Korbonits, MD, PhD, Principal Investigator — Barts and The London
Locations (1):
- Barts and the London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pernicova I, Kelly S, Ajodha S, Sahdev A, Bestwick JP, Gabrovska P, Akanle O, Ajjan R, Kola B, Stadler M, Fraser W, Christ-Crain M, Grossman AB, Pitzalis C, Korbonits M. Metformin to reduce metabolic complications and inflammation in patients on systemic glucocorticoid therapy: a randomised, double-blind, placebo-controlled, proof-of-concept, phase 2 trial. Lancet Diabetes Endocrinol. 2020 Apr;8(4):278-291. doi: 10.1016/S2213-8587(20)30021-8. Epub 2020 Feb 25. PMID 32109422

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were recruited into "Prevention" and "Treatment" algorithms initially. However, only the "Treatment" algorithm proved feasible for logistic reasons. Below are the results relating to patients randomized into the Treatment algorithm.
Groups:
- Metformin: Metformin 850mg TDS for 12 weeks
- Placebo: Placebo 850mg TDS for 12 weeks
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 26 | 27
Abto Keep Appoinment Shedule | 23 | 24
Tolerated at Least 1.7g/Day Dose | 19 | 24
Glucocorticoid Dose as Inc Cri | 19 | 22
Did Not Develop Overt Diabetes | 19 | 21
Completed | 19 | 21
Not Completed | 7 | 6
Not completed — Protocol Violation | 7 | 6

BASELINE CHARACTERISTICS:
Population: Heterogeneous but well matched treatment groups
Groups:
- Metformin: Metformin 850mg TDS
- Placebo: Placebo 850mg TDS
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (15) | 45 (15) | 46 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 27 | 53
  Unknown or Not Reported | 0 | 0 | 0
visceral to subcutanous fat ratio [Median (Inter-Quartile Range); unit: ratio] — Visceral to subcutaneous fat area ratio as assessed by CT at level L4
  ratio | 0.44 [0.33 to 0.67] | 0.58 [0.34 to 0.84] | 0.50 [0.33 to 0.76]
HOMA2-IR [Median (Inter-Quartile Range); unit: HOMA score] — The homeostatic model assessment (HOMA) is a method used to quantify insulin resistance using a HOMA model (https://www.dtu.ox.ac.uk/homacalculator/)
  HOMA score | 4.7 [2.2 to 5.5] | 4.2 [2.8 to 5.4] | 4.4 [2.2 to 5.3]

OUTCOME MEASURES:

1. Primary Outcome: CT Abdomen
Description: change in visceral/subcutaneous fat
Time Frame: 3 months minus baseline
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 19 | 21
ratio | 0.08 (0.19) | -0.03 (0.22)

2. Secondary Outcome: HOMA2-IR
Description: The homeostatic model assessment (HOMA) is a method used to quantify insulin resistance and beta (β)-cell function. HOMA2-IR is a computer model that uses fasting plasma insulin and glucose concentrations to estimate insulin resistance which is the reciprocal of insulin sensitivity (%S)(100/%S) as a percentage of a normal reference population (normal young adults). HOMA2-IR is calculated using the HOMA model: www.dtu.ox.ac.uk/homacalculator/
Time Frame: 3 months minus baseline
Measure: Mean (Standard Deviation); unit: HOMA score
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 19 | 21
HOMA score | 0.22 (3.26) | 2.35 (3.23)

ADVERSE EVENTS:
Time Frame: 6 months
Description: adverse event definition is matching the definition of clinicaltrials.org
Arm/Group | Metformin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/26 | 9/27
Other Adverse Events (participants affected / at risk) | 26/26 | 22/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin (N=26) | Placebo (N=27)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ischaemic heart disease (Cardiac disorders) | 1 | 0
Diverticulitis (Gastrointestinal disorders) | 0 | 1
Atypical chest pain (Cardiac disorders) | 0 | 1
Raynaud's (Vascular disorders) | 0 | 1
Severe osmotic symptoms (Endocrine disorders) | 0 | 2
Exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin (N=26) | Placebo (N=27)
Gastrointestinal side-effects (Gastrointestinal disorders) | 16 | 9
Other (General disorders) | 10 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes